CLINICAL TRIAL: NCT04910035
Title: The Effect of Square Stepping Exercises Training on Lower Extremity Motor Performance, Muscle Strenght and Muscle Quality in Healthy Young People: a Single-Blind, Randomized, Controlled Clinical Trial
Brief Title: The Effect of Square Stepping Exercises Training on Lower Extremity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nigde Omer Halisdemir University (Other)
Collaborators: Pamukkale University (Other)
Responsible Party: Principal Investigator, Asli Demirtaş, Principal Investigator, Nigde Omer Halisdemir University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: (11.06.2019-11)
Record Dates: First submitted 2021-05-04; First posted 2021-06-02 (Actual); Last update posted 2024-09-03 (Actual); Status verified 2021-06

CONDITIONS: Sedentary Healthy Young Individuals
Keywords: Square-stepping exercises; Healthy young individuals; Motor performance; Muscle strength; Muscle quality

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Single (Outcomes Assessor)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Training Group (Active Comparator): Throughout 3 weeks SSE training was administered 4 days a week for a length of 45 minutes in each session. All the analyses were conducted at the start and at the end of 3-week long training.
  Interventions: Other: Exercises Training
- Control Group (No Intervention): This group has no intervention. Evaluations were only made at the start and at the end of 3-week long.

INTERVENTIONS:
Other: Exercises Training — SSE is performed on a thin exercise mat divided into 40 small squares in 250 cm x 100 cm of size (25 cm each part). Participants are given patterns of a few steps and asked to take steps that match them. Participants must, in principal, move ahead in line with the length forward with no contact on the lines forming the squares. Forward, backward, lateral and oblique stepping patterns are required. Stepping patterns get increasingly difficult. Each pattern consists of 2 to 16 steps; participants are asked to repeat step pattern till the end of exercise mat. Upon completing a pattern, another pattern in the same mirror-image is repeated. In essence each pattern is reiterated for 3-5 times and next its mirror-image pattern is repeated but if participants face challenge in performing the pattern it is repeated till the pattern is learnt
  Other Names: Square-steeping exercise
  Arms: Training Group

SUMMARY:
Physical activity plays an indispensable role to lead a healthy life. Square-stepping exercises (SSE) are aerobic exercises.Our study was designed to investigate the effects of square-stepping exercise training on lower-extremity motor performance, muscle strength, and muscle quality of sedentary healthy young individuals.

DETAILED DESCRIPTION:
A total of 120 volunteers within the age range of 20-25 participated in the research. Participants were randomly divided into two groups, as 60 participants were study group (35 females, 25 males) and 60 participants were control group (35 females, 25 males). Demographic data and exercise habit of the individuals were documented. Participants' lower-extremity motor performance was analyzed through Vertical Jumping, Side Jumping, One Leg Squat, and Step-Up tests. Participants' muscle strength was analyzed through Hand-Held Dynamometer. Also, participants' muscle quality was analyzed through Muscle Quality Index. Throughout 3 weeks SSE training was administered 4 days a week for a length of 45 minutes in each session. All the analyses were conducted at the start and at the end of 3-week long training

ELIGIBILITY:
Inclusion Criteria:

* 20-25 years old,
* Not attending any exercise program for the last 1 year,
* Not having a neurological, orthopedic disease or any disease affecting lower extremity,
* Not having any lower-extremity surgery,
* Individuals without vision and/or hearing problems were included in the study.

Exclusion Criteria:

* Having a vision and/or hearing problem,
* Having neurological, psychiatric, and/or orthopedic problems that affect walking,
* Individuals with lower-extremity surgery were excluded from the study.

Ages: 20 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2019-09-10 (Actual); Primary Completion 2020-05-10 (Actual); Study Completion 2020-05-10 (Actual)

PRIMARY OUTCOMES:
Muscle Quality İndex | 3 weeks
  Muscle quality was determined through Muscle Quality Index (MQI) which is a valid and reliable method developed by Takai et al. MQI measures 5 repetition sit-to-stand test duration (sec). MQI is calculated by measuring the 5-repetition sit-to-go test duration (sec), body weight (kg), and leg length (L-m). In the calculation, the formula "(L-0,5)*5*weight*g/5" repetitions sit-to-stand test duration is employed.
Muscle Strength | 3 weeks
  Hand-Held Dynamometer
Motor Performance Assessment 1 | 3 weeks
  Vertical Jumping
Motor Performance Assessment 2 | 3 weeks
  Step-Up
Motor Performance Assessment 3 | 3 weeks
  One Leg Squat
Motor Performance Assessment 4 | 3 weeks
  Side Jumping

CONTACTS AND LOCATIONS:
Locations (1):
- Nigde Omer Halisdemir University, Niğde, Bor, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No